CLINICAL TRIAL: NCT01081600
Title: Imaging the Effect of HSP90 Inhibitor AUY922 on HER2 Expression by Means of 89Zr-trastuzumab PET. Side Study to Phase I-II Study With AUY922 in Either HER2 or ER Positive Locally Advanced or Metastatic Breast Cancer: Protocol CAUY922A2101
Brief Title: 89Zr-trastuzumab PET for Imaging the Effect of HSP90 Inhibition
Acronym: AUY922
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, Principal investigator, University Medical Center Groningen
Other Study IDs: 27112008 version 1; 2008-005751-26 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: Heat shock protein; breast cancer; PET imaging; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — X-Rays; zirconium-89-trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AUY922: Patients with HER2 positive breast cancer which has become trastuzumab resistent.
  Interventions: Other: Imaging with 89Zr-trastuzumab PET

INTERVENTIONS:
Other: Imaging with 89Zr-trastuzumab PET — Injection with 89Zr-trastuzumab and 89Zr-trastuzumab PET scan.
  Other Names: 89Zr-trastuzumab

SUMMARY:
HSP90 inhibition is a potentially new targeted drug modality in the treatment of HER2 positive, trastuzumab refractory breast cancer. Little is known about the pharmacodynamics of HSP90 inhibitors in vivo, but non-invasive PET/CT imaging in a xenograft mouse model could visualize and quantify HER2 reduction after AUY922 treatment by 89Zr-trastuzumab PET imaging. Two doses of 50 mg/kg AUY922 resulted in a decrease in HER2 expression of approximately 50%, quantified 6 days after the last administration of AUY922.

Visualizing HER2 expression in breast cancer patients before and early following HSP90 inhibition by means of 89Zr-trastuzumab PET, is likely to provide insight in the early in vivo effect of HSP90 inhibition and could potentially support patient tailored therapy.

DETAILED DESCRIPTION:
This study is designed as a side study to the multicenter, international phase I-II trial with the HSP90 inhibitor AUY922 (protocol CAUY922A2101), as part of the biomarker assessment. In protocol CAUY922A2101, section 4, the design of this phase I-II trial is described (p36, 37). Briefly, a dose-escalation study is performed according to phase I design. This part is followed by a dose-expansion study according to a phase II design. In the latter part, breast cancer patients are enrolled that are either refractory to hormone- or trastuzumab treatment (both treatment arms, n=40 patients). Patients with HER2 positive, trastuzumab refractory breast cancer, will receive a 89Zr-trastuzumab PET scan as part of the present side study protocol, which will be performed in collaboration with the Royal Marsden Hospital (United Kingdom).

To this end, a 89Zr-trastuzumab PET scan will be performed before (baseline) and during treatment with the HSP90 inhibitor AUY922, as described below.

A minimum of six patients are needed to evaluate whether the 89Zr-trastuzumab PET scan can be used for the detection of a decrease of HER2 expression, induced by HSP90 inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2 positive, trastuzumab (and lapatinib) refractory breast cancer
* Participation in the phase I-II trial with HSP90 inhibitor AUY922 (in- and exclusion criteria for this study with AUY922 are described in protocol CAUY922A2101.

Exclusion Criteria:

* No participation in the phase I-II trial with HSP90 inhibitor AUY922 (CAUY922A2101. Clinical trials no. NCT00526045A)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 positive breast cancer which has become trastuzumab resistent, who are participating in the phase I-II trial with HSP90 inhibitor AUY922
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To show the effect of the HSP90 inhibitor AUY922 on HER2 expression by means of 89Zr-trastuzumab PET scanning. | 2 years
  Primary endpoint: measurement of decreased HER2 expression compared to baseline. A decline is defined as a decrease of at least 30% in mean Standardized Uptake Value (SUV) in a maximum of three lesions.

CONTACTS AND LOCATIONS:
Overall Officials: C.P. Schröder, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands